CLINICAL TRIAL: NCT00824447
Title: A Randomised, DB, Plcb Controlled, Multicentre, Multinat. Phase II/III FU Study to Assess Longterm Efficacy and Safety of 3 Different Dose Regimens of Oralgen® GrassPollen in Patients With Grass Pollen Related Allergic Rhinoconjunctivitis
Brief Title: Long-term Efficacy and Safety Study With Oralgen Grass Pollen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Artu Biologicals (Industry)
Responsible Party: Dr. F.F. Roossien, Artu Biologicals Europe B.V.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB0602/1; 2007-002477-31 (EudraCT Number)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: randomised; double-blind; placebo-controlled; long-term efficacy and safety; Oralgen® Grass Pollen; allergic rhinoconjunctivitis; Allergy; Rhinoconjunctivitis; Immunotherapy; Grass pollen extract
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo control (Placebo Comparator): Placebo control
  Interventions: Other: placebo
- Grass pollen extract, twice weekly (Active Comparator): Grass pollen extract, 9,500 BU, given twice weekly
  Interventions: Drug: Oralgen
- Grass pollen extract daily (Active Comparator): Grass pollen extract, 9,500 BU, given daily
  Interventions: Drug: Oralgen
- Increased dose of grass pollen extract (Active Comparator): Increased dose of grass pollen extract, 19,000 BU, given daily
  Interventions: Drug: Oralgen

INTERVENTIONS:
Drug: Oralgen — allergen solution sublingually
  Other Names: grasspollen extract
  Arms: Grass pollen extract daily; Grass pollen extract, twice weekly; Increased dose of grass pollen extract
Other: placebo — placebo control
  Other Names: Placebo control
  Arms: Placebo control

SUMMARY:
This study is designed to give additional information on the efficacy, safety and local effects (tolerability) of a dose of sublingual immunotherapy administered once a day, during a second grass pollen season.

DETAILED DESCRIPTION:
Allergy is one of the most common chronic diseases. Allergies to grass, weed, and tree pollens characteristically result in seasonal rhinitis symptoms commonly termed hay fever. The risk of developing asthma has been noted to be higher in patients with rhinitis than among the general population (10% versus 3.6%), confirming the fact that rhinitis is often the first step of the natural history of asthma.

Although several drugs effectively manage the symptoms of allergic rhinitis, conjunctivitis or asthma, they do not represent an etiopathogenic treatment of the considered diseases, and do not prevent the reappearance of the symptoms at the end of the treatment.

Immunotherapy is generally considered to be appropriate for patients in whom rhinitis symptoms cannot be controlled by an optimal medication regimen and avoidance of the allergens. At present, specific immunotherapy is the only therapy available that acts on the main cause of the allergic reaction by modifying or down-regulating the immune response.

Allergen immunotherapy is the administration of gradually increasing quantities of an allergen vaccine (extract) to an allergic subject, to reach a maintenance dose, which is effective in reducing the symptoms associated with exposure to the causative allergen.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the in and exclusion criteria for study AB0602 and successfully finished this study.
* Patients who have given their written consent to participate in this study.
* Patients who are willing to comply with the protocol and understand the information given.
* Female patients of childbearing potential are eligible if they are not sexually active or if they use a medically accepted contraceptive method.
* Negative urine pregnancy test if female at the end of the previous study.

Exclusion Criteria:

* Pregnancy, breast-feeding / lactation or sexually active women of childbearing potential who are not using a medically accepted contraceptive method.
* Patients who were non-compliant during study AB0602.
* Patients with a past or current disease, which as judged by the investigator, may affect the patient's participation in or the outcome of this study.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pollen Season Rhinoconjunctivitis Total Symptom Score | site specific pollen season

SECONDARY OUTCOMES:
Rescue medication usage | one year
Proportion of symptom-free days during the pollen season | one year
Rhinoconjunctivitis QoL Questionnaire | one year
Global evaluation of the efficacy by the patient | one year
Local and systemic tolerability and other adverse events, labor | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dyonne van Duren, MD, PhD, Principal Investigator — AMPHA Nijmegen, Toernooiveld 220, 6525EC, Nijmegen, The Netherlands; Knut Schaekel, MD, PhD, Principal Investigator — Universitait Klinikum Carl Gustav Carus, Fetscherstrasse 74, SN 01307, Dresden, Germany; Iveta Kozlovska, MD, PhD, Principal Investigator — Centrum Immunologie a allergologie, Pavla Horova 14, 84108 Bratislava, Slovak Republic
Locations (39):
- Bulgaria (7):
  - MHAT PLovdiv, ENT Clinic, Plovdiv
  - Military Medical Academy, Clinic of ENT, Sofia
  - Military Medical Academy, Sofia
  - 5th MHAT, ENT Clinic, Sofia
  - Ministry of interior-central clinical database, Sofia
  - MHAT Sveta Marina, Varna
  - Military Medical Academy, Varna
- Czechia (9):
  - ORL Soukroma praxe, Brno
  - Fakultni nemocnice Brno, Brno-Bohunice
  - Nemocnice Caslav, Čáslav
  - Alergologicka ordinace, Dobruška
  - Alergologicka ambulance, Jablonec nad Nisou
  - Alergologicka ordinace, Kutná Hora
  - Alergologicka ambulance, Ostrava - Hrabuvka
  - Ambulance plicni a alergologicka, Ostrave - Hrabuvka
  - Alergologicka ambulance Okresni nemocnice Tabor, Tábor
- Germany (6):
  - Berufsgen. kliniken Bergmannsheil, Bochum
  - Univ. klinikum Carl Gustav Carus, Dresden
  - MedicoKIT, Goch
  - Johannes-Gutenberg-Universitat Mainz, Mainz
  - Vital Care, München
  - Privataertz. inst. & Forsh. einrichtung, Wiesbaden
- Hungary (5):
  - Svabhegyi Allami Gyermekgyogyintezet pulmonologia, Budapest
  - Szent Janos Korhaz, Budapest
  - Selye Janos Korhaz, Komárom
  - Karolina Korhaz, Mosomagyarovar
  - Tudogyogyintezet Torokbalint, Törökbálint
- Lithuania (4):
  - Kaunas medical University hospital, Kaunas
  - JSC Seimos gydytojas, Vilnius
  - Vilnius Central Outpatient Clinic, Vilnius
  - Vilnius university hospital, Santariskiu Clinic, Vilnius
- Netherlands (4):
  - Ampha Den Bosch / Regio Brabant, 's-Hertogenbosch
  - Ampha De Bilt, De Bilt
  - Ampha, Hengelo
  - AMPHA Nijmegen, Nijmegen
- Slovakia (4):
  - Centrum imunologie a alergologie s.r.o, Bratislava
  - Amb. klinickey imunologie a allergologie UTaRCH, Poprad
  - Ambulancia klinickej imunologie a alergologie, Trenčín
  - Medcentrum s.r.o., Žilina